CLINICAL TRIAL: NCT03679988
Title: Prevalence of Oral Mucosal Alterations in a Sample of Egyptian Patients With Mucocutaneous Ocular Disorders: A Hospital Based Cross Sectional Study
Brief Title: Prevalence of Oral Mucosal Alterations in Mucocutaneous Ocular Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sherin Alaa Eldin Eisa Elsayed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sherin Alaa Eldin Eisa Elsayed, principle investigator , oral medicine department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MCO oral alterations
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Oral Disease; Muco-Cutaneo-Ocular Syndrome
Keywords: oral health status; oral findings; oral manifestations; patient with mucocutaneous ocular disorders; mucocutaneous ocular disorders
MeSH Terms: conditions — Mouth Diseases; Oral Manifestations

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The patients will be selected from the pool of the Clinics (Rheumatology, Ophthalmology and Dermatology) of Faculty of Medicine and (Diagnostic center and Oral Medicine) of Faculty of Dentistry -Cairo University. For each eligible participant, a full history will be obtained followed by thorough clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with one of the mucocutaneous disorder.
* Patient who will agree to participate in the study.
* Patients who will accept to sign the informed consent.

Exclusion Criteria:

* Patients not physically able to participate in survey or clinical oral examination.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A convenience sample of adult patients diagnosed with mucocutanous oculer disorders attending to Clinics (Rheumatology, Ophthalmology and Dermatology) of Faculty of Medicine and (Diagnostic center and Oral Medicine) of Faculty of Dentistry -Cairo University will be enrolled in the study in a consecutive order.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Identifying and recording oral mucosal alterations | 10 min
  clinical examination according to World Health Organization guidelines

SECONDARY OUTCOMES:
Identifying the oral health-related quality of life: OHIP-14 | 10 min
  using Oral Health Impact Profile-14 (OHIP-14) Slade G. and Spencer A.: Development and evolution of the oral health impact profile.
  Community Dent Health, 11 (1): 3-11, 1994 Response categories for the five-point scale are: "Very often", "Fairly often", "Occasionally", "Hardly ever" and "Never".

IPD SHARING:
Plan to Share IPD: Undecided